CLINICAL TRIAL: NCT07192250
Title: The Thoracolumbar AOSpine Injury Score: Clinical And Radiological Outcomes Of Management Of Fractures Having Scores Of 4 And 5: A Prospective Randomized Trial
Brief Title: Thoracolumbar Burst Fracture Management: Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Hamed Kassem Abdelaal (Other)
Responsible Party: Sponsor-Investigator, Ahmed Hamed Kassem Abdelaal, Dr., Sohag University
Organization: Sohag University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 585/9/444
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Evaluation of the Validity of Thoracolumbar AO Spine Injury Score (TL AOSIS) in A3 and A4 Fractures
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- operative group (Active Comparator)
  Interventions: Procedure: short segment TPF
- conservative group (Active Comparator)
  Interventions: Procedure: conservative management

INTERVENTIONS:
Procedure: short segment TPF — short segment transpedicular screw fixation with one or two screws in fractured vertebra
  Arms: operative group
Procedure: conservative management — brace and bed rest with mobilization as tolerated
  Arms: conservative group

SUMMARY:
Between December 2019 to December 2022, patients presenting to causalty department with TL fracture type A3 and A4 with a TL AOSIS scores of 4 and 5 were randomly managed either by conservative or operative management.

DETAILED DESCRIPTION:
Conservative management group was treated by bed rest and brace for 3 weeks followed by early mobilization. Operative management group received management through Short-segment fixation with one or two screws in fractured vertebra when applicable with posterior spinal fusion. Patients were evaluated both clinically regarding pain (VAS score), disability by Oswestry Disability Index (ODI score) and neurological status. Radiological evaluation included local sagittal spinal alignment, including pre- and post- management Cobb angle and local segment kyphosis. Bony fusion was also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients (age 21-55 years old), TL spine fractures of types A3 and A4 with TL AOSIS score 4 or 5. These include different variables; A4N0, A3N1, A3N2 and A3M1N0.

Exclusion Criteria:

* Osteoporotic fractures and skeletally immature patients, associated comorbidities (e.g. bleeding disorders, rheumatoid arthritis), or any fracture type other than A3 and A4, and significant neurological compromise.

Ages: 21 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Pain score | 6 months
  VAS score
healing | 6 months
  radiological union
deformity | 1 year
  Cobb angle

SECONDARY OUTCOMES:
function | 1 year
  ODI score

CONTACTS AND LOCATIONS:
Overall Officials: mohamed younis, lecturer, Principal Investigator — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Sohag Governorate, Egypt